CLINICAL TRIAL: NCT07297641
Title: Intravascular Imaging-Guided Versus Angiography- Guided Percutaneous Coronary Intervention for Drug-eluting In-stent Restenosis
Brief Title: Intravascular Imaging-Guided Versus Angiography- Guided PCI in Patients With DES-ISR
Status: Recruiting | Type: Observational
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Ye-fei, chief physician, Nanjing First Hospital, Nanjing Medical University
Other Study IDs: KY20241223-KS-02
Record Dates: First submitted 2025-12-09; First posted 2025-12-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: PCI; In-stent Restenosis; Intravascular Imaging Device
Keywords: in-stent restenosis; Intravascular imaging device; percutaneous coronary intervention
MeSH Terms: interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intravascular imaging -guidance: Individuals underwent intravascular imaging -guided PCI for lesions diagnosed with ISR
  Interventions: Procedure: percutaneous coronary intervention
- Angiography-guidance: Individuals underwent angiography-guided PCI for lesions diagnosed with ISR
  Interventions: Procedure: percutaneous coronary intervention

INTERVENTIONS:
Procedure: percutaneous coronary intervention — Percutaneous Coronary Intervention for ISR

SUMMARY:
This study aimed to compare the clinical and angiographic outcomes of patients with DES-ISR who underwent repeat PCI with intravascular imaging or angiographic guidance.

DETAILED DESCRIPTION:
Through early revascularization, percutaneous coronary intervention (PCI) and following pharmacotherapy have improved clinical prognosis among patients with coronary artery disease. However, the presence of stent failure events remained posing long-term risk of adverse cardiac events. Although the utilization of drug-eluting stents (DES), the incidence of in-stent restenosis (ISR) continued to occur at an incidence rate of 1-2% annually. Also, the prognosis of ISR was worse than that in denovo lesions considering its complex mechanisms(stent under-expansion, neointimal hyperplasia or neo-atherosclerosis).Compared with coronary angiography, intravascular imaging(OCT/IVUS) provides detailed anatomical information regarding reference vessel dimensions and lesion characteristics, including severity of diameter stenosis, lesion length, and morphology. Identifying the mechanism of stent failure is paramount because the causative factors will influence the selection of treatment strategy, ultimately impacting the prognosis of the revascularization. However, clinical evidence for the exact benefit of intravascular imaging-guidance for ISR lesions is limited.

Therefore, this study aimed to compare the efficacy and safety of intravascular imaging -guided PCI in patients with ISR.

ELIGIBILITY:
Inclusion Criteria:

(1) Patients with DES-ISR lesions; (2) Life expectancy of at least 1 year; (3) DES-ISR lesions occurring for the first time in native coronary arteries and suitable for re-PCI based on angiographic findings.

Exclusion Criteria:

(1) Bare-metal stent in-stent restenosis (BMS-ISR). (2) Non-DES-ISR lesions. (3) Incomplete clinical and angiographic data. (4) Poor quality of IVUS or angiographic images. (5) Recurrent DES-ISR. (6) Optical coherence tomography (OCT) guidance.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The first-time drug-eluting stent in-stent restenosis (DES-ISR) who underwent repeat percutaneous coronary intervention (re-PCI) under angiographic guidance or combined IVUS guidance.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-11-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
MACE | 3-year
  Major adverse cardiovascular events following PCI

SECONDARY OUTCOMES:
Stent expansion | Intraprocedural
  defined as the final minimal luminal area (MLA) within the treatment segment divided by the average reference vessel area
MSA | Intraprocedural
  minimal stent area

CONTACTS AND LOCATIONS:
Overall Officials: Fei Ye, Principal Investigator — Nanjing First Hospital, Nanjing Medical University, 210006 Nanjing, Jiangsu, China
Locations (1):
- Nanjing First Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No
Due to privacy and ethical limitations, the data generated and analyzed in current study are not publicly available but could be obtained from principal investigator upon the approval of ethics committee

REFERENCES:
- [Result] Wang YF, Xu T, Meng PN, You W, Xu Y, Kong XH, Wu XQ, Wu ZM, Zhao MY, Jia HB, Wang F, Ye F. Optical coherence tomography versus angiography to guide percutaneous coronary intervention in patients with in-stent restenosis: an observational study. Coron Artery Dis. 2025 Mar 1;36(2):108-116. doi: 10.1097/MCA.0000000000001458. Epub 2024 Dec 3. PMID 39620882